CLINICAL TRIAL: NCT06665529
Title: 28-day Mortality Prediction for Critically Ill Patients in the Intensive Care Unit: Physician-nurse vs. Score. A Prospective Observational Study
Brief Title: 28-day Mortality Prediction for Critically Ill Patients in the Intensive Care Unit: Physician-nurse vs. Score
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0232-24-MMC
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Mortality Prediction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 28-day mortality prediction by ICU staff and mortality scores — 28-day mortality prediction by ICU staff (three senior physicians and ICU nurse) and mortality scores (APACHE 2, MPM 2 and MODS).

SUMMARY:
There are several scores for predicting mortality within 28 days in the intensive care unit, including APACHE 2, MPM 2 and MODS. These models for predicting mortality can help intensive care physicians to identify patients at high risk of mortality, thus helping them in the decision regarding their admission to the ICU and the management of their care during hospitalization. However, it is not entirely clear whether these models can predict mortality better than an experienced ICU physician or nurse.

The purpose of the study is to compare the ability of a senior ICU physician and nurse to predict mortality within 28 days in intensive care patients and between the predictive ability of three models for mortality prediction, as well as to investigate what were the parameters that particularly influenced the mortality prediction of the medical and nursing staff.

The study will be performed as a prospective observational study and will include approximately 2000 patients. For each patient admitted to intensive care, the risk of mortality will be calculated according to APACHE 2, MPM 2 and MODS. In addition, an independent evaluation by 3 specialist ICU physicians and an experienced ICU nurse will be carried out. The medical and nursing staff's reasons for the risk provided by them will be presented.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU between 1.1.2025 and 1.1.2027.

Exclusion Criteria:

* Patients who were hospitalized in the ICU for less than 72 hours.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU between 1.1.2025 and 1.1.2027.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality prediction by ICU staff vs. mortality scores | 2 years
  28-day mortality prediction by ICU staff (three senior physicians and ICU nurse) and mortality scores (APACHE 2, MPM 2 and MODS).

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided